CLINICAL TRIAL: NCT05001308
Title: Infectious Mediastinitis Among the Strasbourg Universitary Hospital, a Retrospective Cohort
Brief Title: Infectious Mediastinitis Among the Strasbourg Universitary Hospital
Acronym: MEDIASTINITIS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8262
Record Dates: First submitted 2021-08-06; First posted 2021-08-11 (Actual); Last update posted 2021-12-02 (Actual); Status verified 2021-08

CONDITIONS: Mediastinitis
Keywords: Mediastinitis; Sternitis; Deep Sternal Wound Infection
MeSH Terms: conditions — Mediastinitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Mediastinitis are rare but serious infections, with mortality rates varying from 6 to 30% according to the literature. They are essentially linked to surgical management (cardio-thoracic in particular), but some forms can be spontaneous, after extension of an ENT infectious focus, for example.

Despite their seriousness, there is no strong recommendations to define their management, especially concerning antibiotic therapy and its duration.

The aim of this research is to make a descriptive analysis of the cases of mediastinitis at HUS in recent years, and to study the therapeutic strategy used

ELIGIBILITY:
Inclusion Criteria:

* Major subject (≥18 years old)
* Subject diagnosed with mediastinitis between 01/01/2010 and 31/12/2020
* Subject not having expressed his opposition, after information, to the reuse of his data for the purposes of this research.

Exclusion Criteria:

* Subject having expressed opposition to participate in the study
* Subject under guardianship, curatorship or safeguard of justice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subject diagnosed with mediastinitis between 01/01/2010 and 31/12/2020
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-05 (Estimated); Study Completion 2022-05-31 (Estimated)

PRIMARY OUTCOMES:
Analysis of the cases of mediastinitis and the therapeutic strategy used in recent years at University Hospitals of Strasbourg | Files analysed retrospectively from January 01, 2010 to December 31, 2020 will be examined]

CONTACTS AND LOCATIONS:
Overall Officials: Yvon RUCH, MD, Principal Investigator — Service de maladies infectieuses et tropicales - Hôpitaux Universitaires de Strasbourg
Locations (1):
- Service de maladies infectieuses et tropicales - Hôpitaux Universitaires de Strasbourg, Strasbourg, France